CLINICAL TRIAL: NCT04307784
Title: The Effects of Vitamin D3 Supplementation Alone and in a Combination With Omega-3 on the Association of C-peptide With Glycemic Control; A Randomized Controlled Trial in People With Vitamin D Deficiency
Brief Title: The Effects of Vitamin D3 Alone and in a Combination With Omega-3 on the Association of C-peptide With Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRGS-2014-2015-165-6
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Deficiency; vitamin D3; omega-3 fatty acids; glycated Hemoglubine; C-peptide; Insulin resistance; VD3; A1C; HbA1C
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D3 alone Group (Experimental): Treated with VD3 (50.000 IU/week)
  Interventions: Dietary Supplement: VD3
- Omaga-3 alone Group (Experimental): Treated with (1000 mg) wild salmon and fish oil complex (contains 300 mg of n-3FA) once daily.
  Interventions: Dietary Supplement: Omega-3FA
- Vitamin D3 and Omega-3 Combination, Group (Experimental): Treated with 50.000 IU VD3 per week and 1000 mg wild salmon and fish oil complex (contains 300 mg of n-3FA) once daily.
  Interventions: Dietary Supplement: VD3 and Omega-3FA
- Control Group (Experimental): No intervention was given.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: VD3 — VD3 (50.000 IU/week) for 8 weeks
  Arms: Vitamin D3 alone Group
Dietary Supplement: Omega-3FA — Omaga-3FA (300 mg/day) for 8 weeks
  Arms: Omaga-3 alone Group
Dietary Supplement: VD3 and Omega-3FA — VD3 (50.000 IU/week) and (Omega-3FA 300 mg /day) for 8 weeks
  Arms: Vitamin D3 and Omega-3 Combination, Group
Other: Control — No intervention is given
  Other Names: nothing
  Arms: Control Group

SUMMARY:
The Effects of Vitamin D3 alone and in a combination with omega-3 on the association of C-peptide with glycemic control

DETAILED DESCRIPTION:
The data bout the effects of Vitamin D3 (VD3) alone and as a combination with omega-3 fatty acids (Omega-3FA) on the association between C-peptide (CP) and the glycated hemoglobin (HbA1c) is scarce, conflicting and nothing published in the literature review on the combined effect of VD3 and Omega-3FA as a combination on the association of CP with glycemic control.

This study will be conducted to investigate the effects of (VD3) alone and as a combination with Omega-3FA on the association between CP as an insulin secretion marker, and glycemic control parameters represented by glycated Hemoglobin (HbA1c), on people with vitamin D deficiency (VDD).

This randomized, placebo-controlled trial is designed to test the effects of (50,000 IU VD3/ weekly) and (300mg omega-3FA/daily) separately and as a combination for eight weeks, on the serum levels of CP, 25-hydroxy vitamin D (25OHD) and HbA1c. this study will be carried out during winter on 120 healthy Jordanian males and females with VDD with age range (25-50) years. Fasting serum levels for 25OHD, CP, HbA1c, PTH, Calcium, Phosphate, ALT (Alanine aminotransferase) and Urea were assessed at baseline and at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged (30-64)
* Have a medical diagnosis of VDD

Exclusion Criteria:

* Chronic diseases, such as (osteoporosis, cancer, kidney disease(due to the association between prolonged administration of VD3 and kidney stones formation), an endocrine disorder, thalassemia).
* Documented history of allergic reactions to Omega-3FA supplementations

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of 25-hydroxyvitamin D, C-peptide and HbA1C | 8 weeks
  Concentration

SECONDARY OUTCOMES:
Plasma Concentration of PTH and Calcium | 8 weeks
  Concentration

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-samak, PhD, Principal Investigator — Applied Science Private University (ASU)
Locations (1):
- Applied Science University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underline results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published
Access Criteria: Open access

REFERENCES:
- See also: C-peptide: new findings and therapeutic possibilities. — https://www.ncbi.nlm.nih.gov/pubmed/25648391